CLINICAL TRIAL: NCT06803576
Title: Clinical and Microbiological Parameters of Success Following the Application of Osseointegrated Dental Implants. A 10-year Retrospective Study
Brief Title: Clinical and Microbiological Outcomes of Dental Implants After 10-22 Years of Function
Status: Enrolling by invitation | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Ioannis Vouros, Professor, Aristotle University Of Thessaloniki
Other Study IDs: 458/16-4-2021
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pocket Depth; Attachment Loss; Bone Loss in Jaw
Keywords: dental implants; biologic complications; biomet 3i; Long-term results; prosthetic complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peri-implant sulcular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a least 10 years of loaded implants: Patients from a private periodontal office who have functioning implants for at least 10 years (range 10-22 years)

SUMMARY:
Aim: the aim of this retrospective study is to present long-term data (10+ years of functional loading) on the success and survival of ZimVie (3i) implants. Data from a patient pool of a private periodontal office will be used to reexamine patients with at least 10 years of loading of their dental implants.

Parameters to be examined are bone loss, biologic and prosthetic complications, as well as Patient Reported Outcomes (PROMs) to analyze patient satisfaction with dental implant treatment

DETAILED DESCRIPTION:
Aim: the aim of this study is to present long-term data (10+ years of functional loading) on the success and survival of ZimVie (3i) implants.

Clinical relevance: The successful application of dental implants in replacing missing teeth has been proven since the late 1980's. Over the years a great number of changes in implant designs and implant companies have entered in the dental field of practice. One of the most important questions that have to be addressed is the long-term stability and success of dental implants. While some implant brands have shown reliable long-term stability of their implants, there is still a lack of long-term studies (over 10 years of functional loading) for many implant systems, as it is quite hard to follow-up on patients for such a long time. Therefore, long-term data on implant survival and success is particurarly useful, especially if it is based on private practice patient, thus reflecting the aspects of everyday practice of implantology

Materials and methods: A comprehensive search of patient records from the private practice of the primary investigator (A.B.) was conducted and patients that received dental implant placement from 2001 until 2013 will be asked to participate in the study. After signing the relevant consent forms, all patients that are willing to participate in the study will be examined clinically and radiographically. The following parameters will be examined:

1. Age, sex of patient
2. Relevant medical history
3. Smoking history
4. Compliance to recall appointments
5. Early implant losses
6. Years of prosthetic loading of implants
7. Implant characteristics (length, diameter, surface, cylindrical or root-shaped)
8. Type of prosthesis (single or multiple abutments, cemented or screw-retained)
9. Biological complications (mucositis, peri-implantitis)
10. Prosthetic complications (minor, moderate or severe)
11. History of periodontal disease and treatment prior or after implant placement
12. Prosthetic work performed by specialist or general practitioner
13. Maintenance performed by specialist or general practitioner
14. Relevant ridge augmentation procedures during or before implant placement
15. Clinical measurements (Pocket depth, Attachment loss, Bleeding on probing, presence of Plaque) on six site for every implant (MB, B, DB, ML, L, DL)
16. Samples of the peri-implant sulcular fluid will taken with paper points and measured with Elisa kits to calculate the presence of the following biomarkers: RANKL, OPG, Il-a and TNF-b
17. A radiograph will be taken with the parallel cone technique and compared to baseline xrays after implant placement to measure bone stability
18. A questionnaire will be also provided to all study participants to measure satisfaction following implant therapy Data analysis The main parameter to be examined will be bone loss around an implant over time, as that relates to the definitions of peri-implant mucositis and peri-implantitis. Secondary outcomes will also be examined as pertaining to clinical differences according to the variety of 3i implants that have been used. External vs. internal hex, root-shape vs cylindrical, osseotite vs full osseotite vs nanotite surfaces etc. An number of around 100 patients are expected to be examined for a total of 250 implants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Systemic health or controlled medical conditions
* Periodontal health, either no periodontal disease, or previously treated periodontal disease under a supportive periodontal maintenance (SPT) program
* Smokers were included but encouraged to enter a smoking cessation program
* Patients with bruxism or parafunctional habits were included.

Exclusion Criteria:

* Uncontrolled medical conditions
* Active uncontrolled periodontal disease
* Inability to present for the reevaluation appointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient sample of this study is part of a retrospective evaluation of patients who received treatment with dental implants in a private periodontal practice run by a single specialist Periodontist (A.B.) between 2000 and 2013, with at least 10 years of functional loading of their prosthetic work. A comprehensive chart review revealed 208 potential patients, and an effort will be made to invite all of them for a reevaluation appointment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Marginal Bone loss | 10-22 years
  The amount of vertical bone loss around the mesial and distal surface of an implant, when bone levels at time of placement and at reevaluation were compared

SECONDARY OUTCOMES:
Implant Survival and Success Rates | 10-22 years
  Implant Survival Rate was defined as an implant still in place at the time of reevaluation and Implant Success Rate was defined as an implant with marginal bone loss up to 2 mm
Incidence of peri-implant pathology | 10-22 years
  The percentages of implants that are healthy, have peri-implant mucositis or peri-implantitis

OTHER OUTCOMES:
Patient-Reported Outcome Measures | 10-22 years
  Patients will fill out a questionnaire with 13 targeted questions pertaining to their satisfaction with implant treatment. Patients circled one of the possible answers to each question ("Yes, definitely", "Enough", "Not so", "Definitely not", "Don't know", "No anwswer")

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Vouros, DDS PHD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- School of Dentistry, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make IPD available. It also means that a data dictionary (a description of the variables, or types of data, collected for each individual) will be provided so that the data can be fully interpreted.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start date: July , 2025 End date: December 2025
Access Criteria: Any scientist with an interest in this kind of research

REFERENCES:
- [Background] Amelie Bäumer1,2*, Shirin Toekan3, Daniel Saure4 and Gerd Körner2
- [Background] Carra MC, Blanc-Sylvestre N, Courtet A, Bouchard P. Primordial and primary prevention of peri-implant diseases: A systematic review and meta-analysis. J Clin Periodontol. 2023 Jun;50 Suppl 26:77-112. doi: 10.1111/jcpe.13790. Epub 2023 Mar 6. PMID 36807599
- [Background] Chappuis V, Buser R, Bragger U, Bornstein MM, Salvi GE, Buser D. Long-term outcomes of dental implants with a titanium plasma-sprayed surface: a 20-year prospective case series study in partially edentulous patients. Clin Implant Dent Relat Res. 2013 Dec;15(6):780-90. doi: 10.1111/cid.12056. Epub 2013 Mar 18. PMID 23506385
- [Background] Frisch E, Vach K, Ratka-Krueger P. Impact of supportive implant therapy on peri-implant diseases: A retrospective 7-year study. J Clin Periodontol. 2020 Jan;47(1):101-109. doi: 10.1111/jcpe.13206. Epub 2019 Nov 6. PMID 31599464